CLINICAL TRIAL: NCT04899193
Title: A Phase I, Open-label, Randomized, Three-period, Crossover, Single-center Trial to Assess the Bioequivalence of the Co-administration of 900 IU of Follitropin Alfa (Gonal-f) and 450 IU of Lutropin Alfa (Luveris) Versus the Fixed Combination of 900 IU Follitropin Alfa and 450 IU Lutropin Alfa in Pergoveris, Administered SC as Liquid and FD Formulation, in Pituitary Suppressed Healthy Premenopausal Female Chinese Participants
Brief Title: Pergoveris FD and Liquid China BE Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200061_0012
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Healthy; Pergoveris; Bioequivalence; Infertility
MeSH Terms: conditions — Infertility | interventions — follitropin alfa; Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1: First Reference, Then Test 1, Then Test 2 (Experimental): Participants will receive single dose of Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 1 followed by Test 1 drug (Pergoveris FD) on Day 1 in investigation period 2 followed by Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris
- Sequence 2: First Test 1, Then Test 2, Then Reference (Experimental): Participants will receive single dose of Test 1 drug (Pergoveris FD) on Day 1 in investigation period 1 followed by Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 2 followed by Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris
- Sequence 3: First Test 2, Then Reference, Then Test 1 (Experimental): Participants will receive single dose of Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 1 followed by Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 2 followed by Test 1 drug (Pergoveris FD) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris
- Sequence 4: First Reference, Then Test 2, Then Test 1 (Experimental): Participants will receive single dose of Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 1 followed by Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 2 followed by Test 1 drug (Pergoveris FD) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris
- Sequence 5: First Test 1, Then Reference, Then Test 2 (Experimental): Participants will receive single dose of Test 1 drug (Pergoveris FD) on Day 1 in investigation period 1 followed by Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 2 followed by Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris
- Sequence 6: First Test 2, Then Test 1, Then Reference (Experimental): Participants will receive single dose of Test 2 drug (Pergoveris Liquid) on Day 1 in investigation period 1 followed by Test 1 drug (Pergoveris FD) on Day 1 in investigation period 2 followed by Reference drug (Gonal-f/Luveris injection) on Day 1 in investigation period 3. A washout period of 6 days will be maintained between period 1 and 2 and washout period of 17 days will be maintained between period 2 and 3.
  Interventions: Drug: Pergoveris FD; Drug: Pergoveris Liquid; Drug: Gonal-f; Drug: Luveris

INTERVENTIONS:
Drug: Pergoveris FD — Participants will be administered with 900 IU of recombinant human follicle-stimulating hormone (r-hFSH) and 450 IU of recombinant human luteinizing hormone (r-hLH) freeze-dried powder (Freeze-dried Pergoveris) as subcutaneous injection on Day 1 in investigation period 1 or investigation period 2 or investigation period 3. There will be a washout period of 6 days between investigation period 1 and investigation period 2 and 17 days between investigation period 2 and investigation period 3.
Drug: Pergoveris Liquid — Participants will be administered with 900 IU of r-hFSH and 450 IU of r-hLH solution (Pergoveris Liquid) as subcutaneous injection using disposable pen-injector on Day 1 in investigation period 1 or investigation period 2 or investigation period 3. There will be a washout period of 6 days between investigation period 1 and investigation period 2 and 17 days between investigation period 2 and investigation period 3.
Drug: Gonal-f — Participants will be administered with 900 IU of folitropin alfa (Gonal-f) as subcutaneous injection on Day 1 in investigation period 1 or investigation period 2 or investigation period 3. There will be a washout period of 6 days between investigation period 1 and investigation period 2 and 17 days between investigation period 2 and investigation period 3.
Drug: Luveris — Participants will be administered with 450 IU of lutropin alfa (Luveris) as subcutaneous injection on Day 1 in investigation period 1 or investigation period 2 or investigation period 3. There will be a washout period of 6 days between investigation period 1 and investigation period 2 and 17 days between investigation period 2 and investigation period 3.

SUMMARY:
The main purpose of this study is to assess the bioequivalence (BE) of the fixed combination of follitropin alfa and lutropin alfa in Pergoveris freeze-dried (FD) (Test 1) or in Pergoveris Liquid (Test 2) versus the co-administration of Gonal-f and Luveris (Reference), administered subcutaneously (SC) in pituitary suppressed, healthy premenopausal Chinese female participants, at the doses of 900 international unit (IU) of follitropin alfa and 450 IU lutropin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and ECG, blood pressure (systolic and diastolic) and pulse rate
* Participants who have a negative serum pregnancy test before starting Marvelon and on the days before the Pergoveris or Gonal-f/Luveris dose
* Participants who are taking an oral contraceptive pill (OCP) for at least 1 month prior to Screening and are willing to take the combined oral contraceptive pill (COCP) during the study and to recommence taking their own OCP from Day 55 after the first Pergoveris or Gonal-f/Luveris dosing
* Participants with normal baseline follicle stimulating hormone (FSH) (< 12 IU/L) and estradiol (E2) levels [<= 100 picograms per millilitre (pg/mL)] and showing follicle size <= 11 millimeter (mm)
* Participants who had a normal Thinprep cytologic test (TCT) within the last 1 year before Screening (timeframe to be adjusted based on local routine clinical care). If not performed in routine clinical care, participant must be willing to undergo a cervical smear at Screening
* Participants who have a body weight within >= 45 kilogram (kg) and body mass index within the range 18.5 to 29.9 kilogram per meter square (kg/m^2) (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with any condition that, in the Investigator's opinion, constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
* Participants with clinically significant abnormalities of the genital organs as determined by gynecological examination and Trans Vaginal Ultrasound Scan (TVUS) and based on the Investigator's judgment (example., ovarian tumors, non-functional ovarian cysts, endometrial hyperplasia)
* Participants with polycystic ovaries as defined by at least 1 of the following 2 criteria fulfilled: More than 12 follicles < 10 mm mean diameter in either ovary or at least one ovary of > 10 mL volume
* Participants with ovarian follicle-like structures larger than 11 mm (at Screening)
* Participants with positive result for syphilis, human immunodeficiency virus, hepatitis B surface antigen or hepatitis C Virus
* Participants using drugs that may reduce the effectiveness of COCP (e.g., phenytoin, barbiturates, primidone, carbamazapine, oxcarbazepine, topiramate, felbamate,rifampicin, nelfinavir, ritonavir, griseofulvin, oral ketoconazole, and herbal remedies containing Hypericum perforatum [St. John's Wort])
* Participation in any clinical study within 3 months or 5 half-lives, whichever is longer, prior to Screening or during participation Unsuccessful downregulation, demonstrated by serum luteinising hormone (LH) or FSH levels > 2.0 IU/L or E2 levels > 100 pg/mL the day before Pergoveris or Gonal-f/Luveris administration, or showing follicle size > 11 mm
* Participants vaccinated with any Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-Cov-2) vaccine within 4 weeks before administration of study intervention (Marvelon)
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2021-05-08 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Sampling Time After Administration (AUC0-t, adj) of Follitropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Sampling Time After Administration (AUC0-t, adj) of Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC0-inf,adj) of Follitropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Baseline Adjusted Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC0-inf,adj) of Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Baseline Adjusted Maximum Observed Serum Concentration (Cmax,adj) of Follitropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Baseline Adjusted Maximum Observed Serum Concentration (Cmax,adj) of Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Changes From Baseline in Laboratory Parameters | Baseline up to Day 55
Number of Participants with Clinically Significant Changes From Baseline in Vital Signs | Baseline up to Day 55
Number of Participants with Clinically Significant Changes From Baseline in Electrocardiogram (ECGs) Findings | Baseline up to Day 55
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Baseline up to Day 55
Absolute Value and Change From Baseline in Serum Estradiol Levels | Baseline, Day 14 and 39
Change From Baseline in Follicle Size Assessed by Trans Vaginal Ultrasound Scan | Baseline, Day 8, 14, 22, 39 and 55
Change From Baseline in Follicle Number Assessed by Trans Vaginal Ultrasound Scan | Baseline, Day 8, 14, 22, 39 and 55
Number of Participants With Local Tolerability/Injection Site Reactions (ISRs) | At 5 minutes and 1, 2, 4, 6, 12 and 24 hours post-dose
Time to Reach the Maximum Observed Serum Concentration (Tmax) of Follitropin Alfa and Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Apparent Terminal Half-Life (T1/2) of Follitropin Alfa and Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period
Apparent Terminal Elimination Rate Constant (Lambda z) of Follitropin Alfa and Lutropin Alfa | Pre-dose, 2, 4, 6, 7, 8, 9, 10, 12, 15, 18, 24, 36, 48, 72, 96, 120 and 168 hours post-dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200061_0012
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html